CLINICAL TRIAL: NCT02650765
Title: S100 Biomarker in the Acute Management of Mild Head Injuries
Acronym: S100
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other); Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Teemu Luoto, MD, PhD, A/Prof, Tampere University Hospital
Other Study IDs: R15045
Record Dates: First submitted 2015-12-22; First posted 2016-01-08 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Brain Injury; Head Injury
Keywords: Brain injury; Head injury; Computed tomography; Emergency department
MeSH Terms: conditions — Brain Injuries; Craniocerebral Trauma; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Emergency department:
  - S-S100B
  Storage, -70 degrees celsius freezer:
  * Serum 50 microlitres divided into 8 vials (Eppendorf)
  * Plasma divided into 3 vials (Eppendorf)
  * Whole blood (EDTA)
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Indications for head CT imaging after acute head injury — Indications for head CT imaging after acute head injury as per the Scandinavian guidelines for initial management of minimal, mild and moderate head injuries in adults.

SUMMARY:
A prospective validation study of the "Scandinavian guidelines for initial management of minimal, mild and moderate head injuries in adults". Enrolling a consecutive sample of 1000 adult head injury patients from the emergency department of the Tampere University Hospital (Tampere, Finland). A venous blood sample with S100 analytics (+storage blood) is drawn from every patient. The patients are head CT-scanned according to the SNC guidelines. Outcome assessment (GOSE, MRS, Rivermead PCS Questionnaire) is completed as follows: 1 week, 6 months, 1 year, and 2 years.

DETAILED DESCRIPTION:
A prospective clinical head injury study conducted at the Emergency Department of the Tampere University Hospital, which is situated in Tampere, Finland. The hospital takes care of an catchment area of 524 447 inhabitants both from urban and rural areas. About 100 000 patients are treated in the Emergency department annually.

The study aims to improve the emergency evaluation of patients with an acute head injury, especially a mild head injury. About 80% of head CT scan performed on head injury patients in the Emergency Department of the Tampere University Hospital are negative (= no acute traumatic lesion). There is an urgent need to update the head CT imaging criteria/indications in the context of acute head injury in order to reduce the number of unnecessary scanning. More selective head CT indications result in considerable health care savings and decreased exposure to ionizing radiation, among other benefits.

In this study, the investigators implement the "Scandinavian guidelines for initial management of minimal, mild and moderate head injuries in adults" criteria as part of the emergency care of adults head injury patients. By enrolling a large consecutive sample of patients the investigators are validating this new guideline. Emergency department assessment data is combined with long-term outcome parameters and blood-based biomarkers of neurotrauma.

The main aims of the study are:

1. the validation of the Scandinavian guidelines for initial management of minimal, mild and moderate head injuries in adults
2. the examination of novel blood-based biomarkers of acute brain injury that correlate with the radiological severity of the injury and the long-term outcome

ELIGIBILITY:
Inclusion Criteria:

* Head injury

Exclusion Criteria:

* Age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A consecutive sample of adult patients with an acute head injury whom are treated at the emergency department of the Tampere University Hospital, Tampere, Finland
Sampling Method: Probability Sample
Enrollment: 295 (Actual)
Dates: Start 2015-11; Primary Completion 2021-02 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Non-contrast head CT | 0-72h
  Head CT findings: Intracranial traumatic lesions

SECONDARY OUTCOMES:
Glasgow Outcome Scale Extended | 1 week, 6 months, 1 year, and 2 years
  Glasgow Outcome Scale Extended
Modified Rankin Scale | 1 week, 6 months, 1 year, and 2 years
  Modified Rankin Scale
Rivermead PCS Questionnaire | 1 week, 6 months, 1 year, and 2 years
  Rivermead PCS Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Teemu M Luoto, MD, PhD, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland